CLINICAL TRIAL: NCT00098579
Title: Phase I Trial of Doxorubicin and Alvocidib (Flavopiridol; NCI Supplied Agent, NSC 649890) in the Treatment of Metastatic Sarcoma
Brief Title: Doxorubicin Hydrochloride and Alvocidib in Treating Patients With Metastatic or Recurrent Sarcoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00048; 04-075A; U01CA069856 (NIH); NCT01645488 (obsolete NCT alias)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Gastrointestinal Stromal Tumor; Recurrent Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma | interventions — alvocidib; Doxorubicin

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive doxorubicin hydrochloride IV over 5-10 minutes and alvocidib IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients reaching a cumulative doxorubicin dose of 600 mg/m^2 or experiencing cardiotoxicity may receive alvocidib alone at the discretion of the investigator. Cohorts of 3-6 patients receive escalating doses of alvocidib until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Ten additional patients receive treatment at the MTD. Patients are followed every 3 months for 1 year.
  Interventions: Drug: alvocidib; Drug: doxorubicin hydrochloride

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF

SUMMARY:
This phase I trial is studying the side effects and best dose of alvocidib when given with doxorubicin hydrochloride in treating patients with metastatic or recurrent sarcoma that cannot be removed by surgery. Drugs used in chemotherapy, such as doxorubicin hydrochloride and alvocidib, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Alvocidib may also help doxorubicin hydrochloride work better by making tumor cells more sensitive to the drug. Giving more than one drug may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the maximum tolerated dose of flavopiridol (alvocidib) when administered with a fixed dose of doxorubicin (doxorubicin hydrochloride) in patients with unresectable metastatic or locally recurrent sarcoma.

SECONDARY OBJECTIVES:

I. Determine the clinical pharmacokinetics of this regimen in these patients. II. Determine, preliminarily, the therapeutic activity of this regimen in these patients.

III. Correlate pRb, p53, and p21 protein levels with treatment response and apoptosis in patients treated with this regimen.

IV. Correlate NMR biochemical patterns with response in patients treated with this regimen.

OUTLINE: This is an open-label, dose-escalation study of alvocidib.

Patients receive doxorubicin hydrochloride intravenously (IV) over 5-10 minutes and alvocidib IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients reaching a cumulative doxorubicin dose of 600 mg/m^2 or experiencing cardiotoxicity may receive alvocidib alone at the discretion of the investigator. Cohorts of 3-6 patients receive escalating doses of alvocidib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Ten additional patients receive treatment at the MTD. Patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed soft-tissue sarcoma*

  * Unresectable disease
  * Locally recurrent or metastatic disease
* Disease amenable to biopsy (patients treated at the maximum tolerated dose only)
* No known prior or concurrent brain metastases
* Performance status - Karnofsky 60-100%
* Performance status - ECOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL
* Creatinine clearance ≥ 60 mL/min
* Ejection fraction ≥ 50% by MUGA or echocardiogram
* No uncontrolled hypertension
* No myocardial infarction
* No New York Heart Association class II-IV congestive heart failure
* No unstable angina
* No serious cardiac arrhythmia requiring medication
* No peripheral vascular disease ≥ grade 2 within the past year
* No other clinically significant cardiac disease
* No prior deep vein thrombosis
* No other prior vascular thrombus
* No prior pulmonary embolism
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No symptomatic peripheral neuropathy ≥ grade 2
* No other malignancy within the past 5 years except adequately treated basal cell skin cancer or carcinoma in situ of the cervix

  * Carcinoma in situ not considered a second malignancy
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to study drugs
* No psychiatric illness or social situation that would preclude study compliance
* No ongoing or active infection
* No other uncontrolled illness
* See Chemotherapy
* At least 3 weeks since prior immunotherapy and recovered
* At least 3 weeks since prior chemotherapy (6 weeks for carmustine or mitomycin) and recovered
* No more than 2 prior cytotoxic chemotherapy regimens

  * Peroxisome proliferator-activated receptor (PPAR)-gamma agonists, thalidomide, or targeted therapy (i.e., tyrosine kinase inhibitors including imatinib mesylate, sorafenib, or sunitinib malate) do not count as a prior chemotherapy regimen
* No prior anthracyclines
* At least 3 weeks since prior radiotherapy and recovered
* No prior extensive radiotherapy to bone marrow-producing sites (e.g., radiotherapy to both the pelvis and spine)
* At least a 1 week washout period since prior tyrosine kinase inhibitors or other targeted therapy
* Concurrent low-dose warfarin (1 mg per day) to prevent thrombus of a central line allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-10; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
MTD of alvocidib when given every three weeks in conjunction with doxorubicin hydrochloride | Course 1
  Defined as the dose level immediately preceding the dose where 2 or more patients experienced DLT.

SECONDARY OUTCOMES:
Dose limiting toxicity | Weekly during course 1 at initiation of each course thereafter
  Defined as the occurrence of Grade 4 hematologic toxicity 21 days after treatment, Grade 4 hematologic toxicity lasting 7 days or longer, Grade 3 or 4 non-hematologic toxicity, or any delay in treatment of more than two weeks. Evaluated using the National Cancer Institute (NCI) Common Toxicity Criteria. Graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Clinical pharmacokinetics of the regimen | Week 1
  Biopsies will be performed by Tru-Cut or CT guidance. The material obtained will be examined for p21, p53 and pRb expression by immunohistochemistry (IHC) as well as measurements of apoptosis by terminal deoxynucleotidyl transferase (TdT)- mediated dUTP nick end labeling (TUNEL).
Therapeutic activity of alvocidib in combination with doxorubicin hydrochloride in patients with advanced solid tumors | Every 2 courses for the first 6 courses and every 3 courses thereafter
  Evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.

CONTACTS AND LOCATIONS:
Overall Officials: David D'Adamo, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States